CLINICAL TRIAL: NCT04367649
Title: Evaluation of Hall Technique and Atraumatic Restorative Treatment for Management of Caries in the Primary Dentition (A Randomized Controlled Clinical Trial)
Brief Title: Evaluation of Hall Technique and Atraumatic Restorative Treatment for Management of Caries in the Primary Dentition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Dental Public Health clinical instructor and statistician, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hall technique for management
Record Dates: First submitted 2020-04-25; First posted 2020-04-29 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Primary Dental Caries
MeSH Terms: interventions — Dental Atraumatic Restorative Treatment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hall technique (Experimental)
  Interventions: Other: Hall technique
- Atraumatic restorative treatment (Active Comparator)
  Interventions: Other: Atraumatic restorative treatment
- Conventional restorative treatment (Sham Comparator)
  Interventions: Other: Conventional restorative treatment

INTERVENTIONS:
Other: Hall technique — * Orthodontic separators will be used to create space for fitting the stainless crown, then removed after 3-5 days
  * Occlusion will be measured assessing the patient's occlusal-vertical dimensions (OVD) using a modified version of van der Zee and van Amerongen method with a millimeter probe measuring the distance from the lowest point of the gingiva, around the lower canine on the vestibular side up to the point where the tip of the upper canine ends in order to assess the degree of overbite after mounting of the crown.
  * The correct crown size will be selected. The crown should cover all the cusps and approaches the contact points, with a slight feeling of "spring back." till reaching the gingival margin. Cementation will be done using glass ionomer cement
  Arms: Hall technique
Other: Atraumatic restorative treatment — Caries removal using excavators, then restoration using glass ionomer (GIC)
  Arms: Atraumatic restorative treatment
Other: Conventional restorative treatment — Complete caries removal using high-speed hand piece, and an excavator to clear carious dentin from the pulpal wall. Then, stainless steel crown preparation, selection of the proper size with the smallest crown size that completely covers the preparation chosen. The correct occlusogingival crown length will be established. Cementation will be done using glass ionomer cement
  Arms: Conventional restorative treatment

SUMMARY:
The aim of the present study is to evaluate both Hall technique and atraumatic restorative technique in comparison to the conventional restorative technique in the management of carious lesions in primary molars.

DETAILED DESCRIPTION:
This study is a three arm randomized controlled clinical trial. Eligible children will be selected from the outpatient clinic of Pediatric Dentistry and Public Health Department, Faculty of Dentistry, Alexandria University after securing necessary consents. One hundred and fifty five teeth will be randomly allocated into 3 groups fifty two each. Group I will be assigned to Hall technique Group II will be assigned to atraumatic restorative treatment using Glass ionomer cement, and Group III will be assigned to a conventional restoration and will serve as a control.

ELIGIBILITY:
Inclusion Criteria:

* Children free of any systemic disease or special health care needs.
* Cooperative children ( positive/ definitely positive) according to Frankl's behavior rating scale.
* Children who are willing to participate in the study
* Tooth inclusion criteria:

  * Primary molar teeth with occlusal or occlusoproximal carious lesions into dentin (International Caries Detection and Assessment System) (ICDAS) codes: 3-5
  * Absence of clinical signs or symptoms of irreversible pulpitis
  * Absence of fistula or abscess near the selected tooth clinically and radiographically
  * Absence of spontaneous pain
  * Absence of pulp exposure
  * Absence of pathological mobility by placing the points of a pair of tweezers in an occlusal fossa, and gently rocking the tooth bucco-lingually.

Exclusion Criteria:

* Clinical signs and symptoms of irreversible pulpilitis.
* Tooth mobility
* Spontaneous pain

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 155 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Success of the crown (for Hall and conventional techniques) | 1 week
  The presence of a satisfactory crown will be checked. Loss of the crown, perforated crown or restoration fracture are considered failures.
Success of the crown (for Hall and conventional techniques) | 1 month
  The presence of a satisfactory crown will be checked. Loss of the crown, perforated crown or restoration fracture are considered failures.
Success of the crown (for Hall and conventional techniques) | 6 months
  The presence of a satisfactory crown will be checked. Loss of the crown, perforated crown or restoration fracture are considered failures.
Success of the crown (for Hall and conventional techniques) | 12 months
  The presence of a satisfactory crown will be checked. Loss of the crown, perforated crown or restoration fracture are considered failures.
Success of the atraumatic restorative technique | 1 week
  Scoring of the restoration between 0-9. 0: Present, satisfactory. 1: Present, slight deficiency at cavity margin of less than 0.5 mm. 2: Present, slight deficiency at cavity margin of 0.5 mm or more. 3: Present, fracture in restoration. 4: Present, fracture in tooth. 5: Present, overextension of approximal margin of 0.5 mm or more. 6: Not present, most or all of restoration missing. 7: Not present, other restorative treatment performed. 8: Not present, tooth is not present. 9: Unable to diagnose. Success scores are 0 and 1, while failure scores are 2-8.
Success of the atraumatic restorative technique | 1 month
  Scoring of the restoration between 0-9. 0: Present, satisfactory. 1: Present, slight deficiency at cavity margin of less than 0.5 mm. 2: Present, slight deficiency at cavity margin of 0.5 mm or more. 3: Present, fracture in restoration. 4: Present, fracture in tooth. 5: Present, overextension of approximal margin of 0.5 mm or more. 6: Not present, most or all of restoration missing. 7: Not present, other restorative treatment performed. 8: Not present, tooth is not present. 9: Unable to diagnose. Success scores are 0 and 1, while failure scores are 2-8.
Success of the atraumatic restorative technique | 6 months
  Scoring of the restoration between 0-9. 0: Present, satisfactory. 1: Present, slight deficiency at cavity margin of less than 0.5 mm. 2: Present, slight deficiency at cavity margin of 0.5 mm or more. 3: Present, fracture in restoration. 4: Present, fracture in tooth. 5: Present, overextension of approximal margin of 0.5 mm or more. 6: Not present, most or all of restoration missing. 7: Not present, other restorative treatment performed. 8: Not present, tooth is not present. 9: Unable to diagnose. Success scores are 0 and 1, while failure scores are 2-8.
Success of the atraumatic restorative technique | 12 months
  Scoring of the restoration between 0-9. 0: Present, satisfactory. 1: Present, slight deficiency at cavity margin of less than 0.5 mm. 2: Present, slight deficiency at cavity margin of 0.5 mm or more. 3: Present, fracture in restoration. 4: Present, fracture in tooth. 5: Present, overextension of approximal margin of 0.5 mm or more. 6: Not present, most or all of restoration missing. 7: Not present, other restorative treatment performed. 8: Not present, tooth is not present. 9: Unable to diagnose. Success scores are 0 and 1, while failure scores are 2-8.
Treatment (restoration) survival | 1 week
  ART restorations, Hall technique and conventional restorations will be scored as satisfactory will be considered "successful," while those presented minor and/or major failures will be considered as "failed."
Treatment (restoration) survival | 1 month
  ART restorations, Hall technique and conventional restorations will be scored as satisfactory will be considered "successful," while those presented minor and/or major failures will be considered as "failed."
Treatment (restoration) survival | 6 months
  ART restorations, Hall technique and conventional restorations will be scored as satisfactory will be considered "successful," while those presented minor and/or major failures will be considered as "failed."
Treatment (restoration) survival | 12 months
  ART restorations, Hall technique and conventional restorations will be scored as satisfactory will be considered "successful," while those presented minor and/or major failures will be considered as "failed."
Radiographic evaluation of the treatment | 6 months
  Digital postoperative periapical radiographs will be obtained using a paralleling device to allow for exact and reproducible alignment of the dental film and the X-ray tube at the different follow up intervals. Teeth will be considered radiographically successful if they showed no evidence of radicular radiolucency, internal or external root resorption or periodontal ligament space widening
Radiographic evaluation of the treatment | 12 months
  Digital postoperative periapical radiographs will be obtained using a paralleling device to allow for exact and reproducible alignment of the dental film and the X-ray tube at the different follow up intervals. Teeth will be considered radiographically successful if they showed no evidence of radicular radiolucency, internal or external root resorption or periodontal ligament space widening

SECONDARY OUTCOMES:
Child satisfaction | immediately after completion of the dental treatment procedures
  The patient's perception of the treatment was assessed by using a faces scale modified to represent satisfaction, indifference, or dissatisfaction . A few minutes will be spent before each procedure to establish rapport with the child and to obtain some notion of the child's understanding of the meaning of those schematic facial expressions. After treatment, the child will be instructed to choose the face that best represented how he/she felt during the procedure.
Assessment of oral cleanliness (plaque) | 1 week
  using plaque index of Sillness and Loe. 0: No plaque. 1: A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface. 2: Moderate accumulation of soft deposits within the gingival pocket, or the tooth and gingival margin which can be seen by the naked eye. 3: Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
Assessment of oral cleanliness (plaque) | 1 month
  using plaque index of Sillness and Loe. 0: No plaque. 1: A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface. 2: Moderate accumulation of soft deposits within the gingival pocket, or the tooth and gingival margin which can be seen by the naked eye. 3: Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
Assessment of oral cleanliness (plaque) | 6 months
  using plaque index of Sillness and Loe. 0: No plaque. 1: A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface. 2: Moderate accumulation of soft deposits within the gingival pocket, or the tooth and gingival margin which can be seen by the naked eye. 3: Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
Assessment of oral cleanliness (plaque) | 12 months
  using plaque index of Sillness and Loe. 0: No plaque. 1: A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface. 2: Moderate accumulation of soft deposits within the gingival pocket, or the tooth and gingival margin which can be seen by the naked eye. 3: Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
Assessment of the gingival condition | 1 week
  using gingival index of Loe and Sillness. 0: Normal gingival. 1: Mild inflammation; slight change in color and slight edema, no bleeding on probing. 2: Moderate inflammation; redness, edema, glazing and bleeding on probing. 3: Severe inflammation; marked redness, edema, ulcerations and tendency towards spontaneous bleeding.
Assessment of the gingival condition | 1 month
  using gingival index of Loe and Sillness. 0: Normal gingival. 1: Mild inflammation; slight change in color and slight edema, no bleeding on probing. 2: Moderate inflammation; redness, edema, glazing and bleeding on probing. 3: Severe inflammation; marked redness, edema, ulcerations and tendency towards spontaneous bleeding.
Assessment of the gingival condition | 6 months
  using gingival index of Loe and Sillness. 0: Normal gingival. 1: Mild inflammation; slight change in color and slight edema, no bleeding on probing. 2: Moderate inflammation; redness, edema, glazing and bleeding on probing. 3: Severe inflammation; marked redness, edema, ulcerations and tendency towards spontaneous bleeding.
Assessment of the gingival condition | 12 months
  using gingival index of Loe and Sillness. 0: Normal gingival. 1: Mild inflammation; slight change in color and slight edema, no bleeding on probing. 2: Moderate inflammation; redness, edema, glazing and bleeding on probing. 3: Severe inflammation; marked redness, edema, ulcerations and tendency towards spontaneous bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Dina Sharaf, M.Sc, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Karin ML Dowidar, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Laila M El Habashy, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Santamaria RM, Innes NP, Machiulskiene V, Evans DJ, Splieth CH. Caries management strategies for primary molars: 1-yr randomized control trial results. J Dent Res. 2014 Nov;93(11):1062-9. doi: 10.1177/0022034514550717. Epub 2014 Sep 12. PMID 25216660
- [Background] Gruythuysen RJ, van Strijp AJ, van Palestein Helderman WH, Frankenmolen FW. [Non-restorative treatment of cavities in temporary dentition: effective and child-friendly]. Ned Tijdschr Geneeskd. 2011;155(42):A3489. Dutch. PMID 22027459
- [Background] Innes NP, Stirrups DR, Evans DJ, Hall N, Leggate M. A novel technique using preformed metal crowns for managing carious primary molars in general practice - a retrospective analysis. Br Dent J. 2006 Apr 22;200(8):451-4; discussion 444. doi: 10.1038/sj.bdj.4813466. PMID 16703041
- [Background] Santamaria RM, Innes NP, Machiulskiene V, Evans DJ, Alkilzy M, Splieth CH. Acceptability of different caries management methods for primary molars in a RCT. Int J Paediatr Dent. 2015 Jan;25(1):9-17. doi: 10.1111/ipd.12097. Epub 2014 Mar 7. PMID 24602167
- [Background] Frencken JE, Holmgren CJ. Caries management through the Atraumatic Restorative Treatment (ART) approach and glass-ionomers: update 2013. Braz Oral Res. 2014;28:5-8. doi: 10.1590/S1806-83242013000600001. No abstract available. PMID 24402057
- [Background] Innes N, Stewart M, Souster G, Evans D. The Hall Technique; retrospective case-note follow-up of 5-year RCT. Br Dent J. 2015 Oct 23;219(8):395-400. doi: 10.1038/sj.bdj.2015.816. PMID 26494348
- [Background] Innes NP, Evans DJ, Stirrups DR. The Hall Technique; a randomized controlled clinical trial of a novel method of managing carious primary molars in general dental practice: acceptability of the technique and outcomes at 23 months. BMC Oral Health. 2007 Dec 20;7:18. doi: 10.1186/1472-6831-7-18. PMID 18096042
- [Background] Innes N, Evans D, Hall N. The Hall Technique for managing carious primary molars. Dent Update. 2009 Oct;36(8):472-4, 477-8. doi: 10.12968/denu.2009.36.8.472. PMID 19927456
- [Background] van der Zee V, van Amerongen WE. Short communication: Influence of preformed metal crowns (Hall technique) on the occlusal vertical dimension in the primary dentition. Eur Arch Paediatr Dent. 2010 Oct;11(5):225-7. doi: 10.1007/BF03262751. PMID 20932395
- [Background] Frencken JE, Pilot T, Songpaisan Y, Phantumvanit P. Atraumatic restorative treatment (ART): rationale, technique, and development. J Public Health Dent. 1996;56(3 Spec No):135-40; discussion 161-3. doi: 10.1111/j.1752-7325.1996.tb02423.x. PMID 8915958
- [Background] Farag A, van der Sanden WJ, Abdelwahab H, Frencken JE. Survival of ART restorations assessed using selected FDI and modified ART restoration criteria. Clin Oral Investig. 2011 Jun;15(3):409-15. doi: 10.1007/s00784-010-0403-0. Epub 2010 Apr 7. PMID 20372951